CLINICAL TRIAL: NCT02949128
Title: Single Arm Study of ALXN1210 in Complement Inhibitor Treatment-naïve Adult and Adolescent Patients With Atypical Hemolytic Uremic Syndrome (aHUS)
Brief Title: Study of ALXN1210 in Complement Inhibitor Treatment-Naïve Adult and Adolescent Participants With Atypical Hemolytic Uremic Syndrome (aHUS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALXN1210-aHUS-311; 2016-002027-29 (EudraCT Number)
Record Dates: First submitted 2016-10-25; First posted 2016-10-31 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Atypical Hemolytic Uremic Syndrome (aHUS)
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome | interventions — ravulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ravulizumab (Experimental): Participants were administered weight-based doses of ravulizumab every 8 weeks for 26 weeks in the Initial Evaluation Period.
  After the Initial Evaluation Period, participants could enter an Extension Period and receive ravulizumab until the product registration or approval (in accordance with country-specific regulations) or for up to 4.5 years, whichever occurs first.
  Interventions: Biological: Ravulizumab

INTERVENTIONS:
Biological: Ravulizumab — Single loading dose on Day 1, followed by regular maintenance dosing beginning on Day 15, based on weight: ≥ 40 to < 60 kilograms (kg), 2400 milligrams (mg) loading, then 3000 mg every 8 weeks; ≥ 60 to < 100 kg, 2700 mg loading, then 3300 mg every 8 weeks; ≥ 100 kg, 3000 mg loading, then 3600 mg every 8 weeks.
  Other Names: ALXN1210; Ultomiris

SUMMARY:
The purpose of the study is to assess the safety and efficacy of ravulizumab to control disease activity in adolescent and adult participants with aHUS who had not previously used a complement inhibitor.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 12 years of age and weighing ≥ 40 kg at the time of consent.
2. Evidence of thrombotic microangiopathy, including low platelet count, hemolysis (breaking of red blood cells inside of blood vessels), and decreased kidney function.
3. Documented meningococcal vaccination not more than 3 years prior to, or at the time of, initiating study drug. Participants who received a meningococcal vaccine less than 2 weeks before initiating ravulizumab treatment must have received treatment with appropriate prophylactic antibiotics until 2 weeks after vaccination. Participants who had not been vaccinated prior to initiating ravulizumab treatment should have received prophylactic antibiotics prior to and for at least 2 weeks after meningococcal vaccination. Participants < 18 years of age must have been vaccinated against haemophilus influenzae type b and streptococcus pneumoniae according to national and local vaccination schedule guidelines.
4. Female participants of childbearing potential and male participants with female partners of childbearing potential had to use highly effective contraception starting at screening and continuing until at least 8 months after the last dose of ravulizumab.

Exclusion Criteria:

1. A disintegrin and metalloproteinase with a thrombospondin type 1 motif, member 13 deficiency (activity < 5%).
2. Shiga toxin-related hemolytic uremic syndrome.
3. Positive direct Coombs test.
4. Pregnancy or breastfeeding.
5. Identified drug exposure-related hemolytic uremic syndrome (HUS).
6. Bone marrow transplant/hematopoietic stem cell transplant within last 6 months prior to start of Screening.
7. HUS related to known genetic defects of cobalamin C metabolism.
8. Systemic sclerosis (scleroderma), systemic lupus erythematosus, or antiphospholipid antibody positivity or syndrome.
9. Chronic dialysis (defined as dialysis on a regular basis as renal replacement therapy for end-stage kidney disease).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (4):
  - Clinical Trial Site, Fort Wayne, Indiana
  - Clinical Trial Site, Durham, North Carolina
  - Clinical Trial Site, Winston-Salem, North Carolina
  - Clinical Trial Site, Columbus, Ohio
- Australia (3):
  - Clinical Trial Site, Clayton
  - Clinical Trial Site, Geelong
  - Clinical Trial Site, Parkville
- Clinical Trial Site, Vienna, Austria
- Clinical Trial Site, Brussels, Belgium
- Clinical Trial Site, London, Canada
- France (6):
  - Clinical Trial Site, Bordeaux
  - Clinical Trial Site, Clermont-Ferrand
  - Clinical Trial Site, Lille
  - Clinical Trial Site, Montpellier
  - Clinical Trial Site, Nice
  - Clinical Trial Site, Paris
- Germany (5):
  - Clinical Trial Site, Aachen
  - Clinical Trial Site, Essen
  - Clinical Trial Site, Hanover
  - Clinical Trial Site, München
  - Clinical Trial Site, Tübingen
- Italy (2):
  - Clinical Trial Site, Bologna
  - Clinical Trial Site, Florence
- Japan (2):
  - Clinical Trial Site, Saitama
  - Clinical Trial Site, Tokyo
- Russia (2):
  - Clinical Trial Site, Moscow
  - Clinical Trial Site, Saint Petersburg
- South Korea (2):
  - Clinical Trial Site, Gyeonggi-do
  - Clinical Trial Site, Seoul
- Spain (3):
  - Clinical Trial Site, Barcelona
  - Clinical Trial Site, Madrid
  - Clinical Trial Site, Valencia
- Taiwan (2):
  - Clinical Trial Site, Taichung
  - Clinical Trial Site, Taipei
- United Kingdom (2):
  - Clinical Trial Site, Cardiff
  - Clinical Trial Site, London

REFERENCES:
- [Result] Barbour T, Scully M, Ariceta G, Cataland S, Garlo K, Heyne N, Luque Y, Menne J, Miyakawa Y, Yoon SS, Kavanagh D; 311 Study Group Members. Long-Term Efficacy and Safety of the Long-Acting Complement C5 Inhibitor Ravulizumab for the Treatment of Atypical Hemolytic Uremic Syndrome in Adults. Kidney Int Rep. 2021 Mar 24;6(6):1603-1613. doi: 10.1016/j.ekir.2021.03.884. eCollection 2021 Jun. PMID 34169200
- [Derived] Matsumoto M, Shimono A, Yokosawa J, Hirose K, Wang E, Maruyama S. Correlation between a 2-week change in platelet count and clinical outcomes after the initiation of ravulizumab treatment in adult patients with atypical hemolytic uremic syndrome: post-hoc analysis of the phase III trial. Thromb J. 2024 Oct 28;22(1):93. doi: 10.1186/s12959-024-00652-1. PMID 39468592
- [Derived] Cammett TJ, Garlo K, Millman EE, Rice K, Toste CM, Faas SJ. Exploratory Prognostic Biomarkers of Complement-Mediated Thrombotic Microangiopathy (CM-TMA) in Adults with Atypical Hemolytic Uremic Syndrome (aHUS): Analysis of a Phase III Study of Ravulizumab. Mol Diagn Ther. 2023 Jan;27(1):61-74. doi: 10.1007/s40291-022-00620-3. Epub 2022 Nov 4. PMID 36329366
- [Derived] Pugh D, O'Sullivan ED, Duthie FA, Masson P, Kavanagh D. Interventions for atypical haemolytic uraemic syndrome. Cochrane Database Syst Rev. 2021 Mar 23;3(3):CD012862. doi: 10.1002/14651858.CD012862.pub2. PMID 33783815
- [Derived] Gackler A, Schonermarck U, Dobronravov V, La Manna G, Denker A, Liu P, Vinogradova M, Yoon SS, Praga M. Efficacy and safety of the long-acting C5 inhibitor ravulizumab in patients with atypical hemolytic uremic syndrome triggered by pregnancy: a subgroup analysis. BMC Nephrol. 2021 Jan 6;22(1):5. doi: 10.1186/s12882-020-02190-0. PMID 33407224

RESULTS

PARTICIPANT FLOW:
Groups:
- Ravulizumab: Participants received weight-based dosages of ravulizumab for 26 weeks during the Initial Evaluation Period. Participants received a loading dose of ravulizumab intravenously on Day 1, followed by maintenance dosing on Day 15 and once every 8 weeks thereafter. After the Initial Evaluation Period, participants entered an Extension Period and received ravulizumab until the product registration or approval (in accordance with country-specific regulations) or for up to 4.5 years, whichever occurs first.
Period: Initial Evaluation Period (26 Weeks)
Arm/Group | Ravulizumab
Started | 58
Received At Least 1 Dose of Study Drug | 58
Completed (Completed the Initial Evaluation Period) | 49
Not Completed | 9
Not completed — Failed to Meet Eligibility Criteria | 2
Not completed — Adverse Event | 3
Not completed — Death | 2
Not completed — Physician Decision | 1
Not completed — Protocol Violation | 1
Period: Extension Period (Up to 4.5 Years)
Arm/Group | Ravulizumab
Started | 49
Received At Least 1 Dose of Study Drug | 47
Completed | 28
Not Completed | 21
Not completed — Death | 1
Not completed — Physician Decision | 5
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 9
Not completed — Other than specified | 5

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of ravulizumab, had at least 1 post-baseline efficacy assessment, and met pre-specified eligibility criteria.
Arm/Group | Ravulizumab
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (14.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 29
  More than one race | 0
  Unknown or Not Reported | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage Of Participants With Complete Thrombotic Microangiopathy (TMA) Response at Week 26
Description: Complete TMA response during the 26-week Initial Evaluation Period is a composite outcome measure that required normalization of hematological parameters (platelet count and lactate dehydrogenase [LDH]) and improvement in kidney function (≥25% reduction in serum creatinine from baseline); for participants on dialysis, baseline was established at least 6 days after the end of dialysis. Participants had to meet these criteria for 2 separate assessments obtained at least 4 weeks (28 days) apart, and any measurement in between. To be considered a responder during the 26-week Initial Evaluation Period, the latest time point a participant could first meet the response criteria was 28 days before the Week 26 (Day 183) assessment. Formal statistical comparison analyses were not planned for this study. The percentage was based on the responders among treated participants. The 95% confidence interval (CI) was based on the asymptotic Gaussian approximation method with a continuity correction.
Time Frame: Week 26
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Ravulizumab: Participants received weight-based dosages of ravulizumab for 26 weeks during the Initial Evaluation Period. Participants received a loading dose of ravulizumab intravenously on Day 1, followed by maintenance dosing on Day 15 and once every 8 weeks thereafter.
Arm/Group | Ravulizumab
Number analyzed (Participants) | 56
percentage of participants
  Complete TMA Response | 53.6 [39.6 to 67.5]
  Platelet count normalization | 83.9 [73.4 to 94.4]
  LDH normalization | 76.8 [64.8 to 88.7]
  ≥ 25% improvement in serum creatinine from baseline | 58.9 [45.2 to 72.7]

2. Secondary Outcome: Time To Complete TMA Response
Description: Participants that did not have a response were censored at the date of last visit or study discontinuation at the time when the analysis was performed. The time to complete TMA Response is reported in days. The time of the event of a confirmed complete TMA response was considered the first time point at which all the criteria for complete TMA response were met.
Time Frame: Baseline through Week 114
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Ravulizumab
Number analyzed (Participants) | 56
days | 86.0 [42.0 to NA] — Participants who did not have a response were censored at the date of last visit or study discontinuation.

3. Secondary Outcome: Participants Who Do Not Require Dialysis at Weeks 26 and 52
Description: For participants requiring dialysis within 5 days prior to ALXN1210 treatment initiation, the number of participants no longer requiring dialysis is reported
Time Frame: Week 26 and Week 52
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of ravulizumab, had at least 1 post-baseline efficacy assessment, met pre-specified eligibility criteria, and had evaluable data at specified timepoint. Here, Overall Number of Participants analyzed signifies those who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Ravulizumab
Number analyzed (Participants) | 24
Participants
  Week 26 | 16
  Week 52: number analyzed (Participants) | 22
  Week 52 | 16

4. Secondary Outcome: Proportion Of Participants With Complete TMA Response At Week 52
Description: The proportion of participants considered responders, along with a 2-sided 95% CI for the Week 52 time point, is reported. To be considered a responder during the 26-week Initial Evaluation Period, the latest time point a participant could first meet the response criteria was 28 days before the Week 26 (Day 183) assessment (components of the response maintained for at least 28 days).
Time Frame: Week 52
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of ravulizumab, had at least 1 post-baseline efficacy assessment, met pre-specified eligibility criteria, and had evaluable data at specified timepoint (Week 52).
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Ravulizumab
Number analyzed (Participants) | 44
proportion of participants
  Complete TMA Response | 0.500 [0.346 to 0.654]
  Platelet Count Normalization | 0.909 [0.783 to 0.975]
  LDH Normalization | 0.750 [0.597 to 0.868]
  ≥25% improvement in serum creatinine from baseline | 0.659 [0.501 to 0.795]

5. Secondary Outcome: Change From Baseline In Estimated Glomerular Filtration Rate (eGFR) At Weeks 26 and 52
Description: Kidney function evaluated by eGFR was summarized at baseline and the Week 26 and Week 52 time points using descriptive statistics for continuous variables for the observed value, as well as the change from baseline. The baseline value was defined as the average of the values from the assessments performed prior to the first study drug infusion (these could include results from Screening and the Day 1 visit). A value of 10 milliliters (mL)/minute (min)/1.73 meters squared (m^2) for eGFR was imputed for participants requiring dialysis for acute kidney injury. The observed value and change from baseline are reported in mL/min/1.73 m^2. An increase indicated improvement in kidney function.
Time Frame: Baseline, Week 26 and Week 52
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of ravulizumab, had at least 1 post-baseline efficacy assessment, met pre-specified eligibility criteria, and had evaluable data at the specified timepoint (Week 26 or Week 52).
Measure: Median (Full Range); unit: mL/min/1.73 m^2
Arm/Group | Ravulizumab
Number analyzed (Participants) | 48
mL/min/1.73 m^2
  Baseline | 10.00 [4 to 80]
  Change From Baseline at Week 26: number analyzed (Participants) | 47
  Change From Baseline at Week 26 | 29.00 [-13 to 108]
  Change From Baseline at Week 52: number analyzed (Participants) | 43
  Change From Baseline at Week 52 | 23.00 [-13 to 95]

6. Secondary Outcome: Participants With Change From Baseline In CKD Stage At Weeks 26 and 52
Description: The CKD stage is presented as the change from baseline in the participants that Improved (excluding those with Stage 1 [normal renal function] at baseline as they cannot improve), Worsened (excluding those with Stage 5 at baseline as they cannot worsen), and Stayed the Same, compared to the CKD stage at baseline. Baseline was derived based on the last available eGFR before starting treatment. Stage 5 was considered the worst category, while Stage 1 was considered the best category. A 2-sided 95% CI for the proportion, based on exact confidence limits using the Clopper-Pearson method, was provided for each category. The CKD stage was classified based on the National Kidney Foundation Chronic Kidney Disease Stage.
Time Frame: Baseline, Week 26, and Week 52
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of ravulizumab, had at least 1 post-baseline efficacy assessment, met pre-specified eligibility criteria, and had evaluable data at the specified timepoint (Week 26 or Week 52). Here, Overall 'Number of Participants Analyzed' signifies those who were evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Ravulizumab
Number analyzed (Participants) | 47
Participants
  Week 26, Improved | 32
  Week 26, Worsened | 2
  Week 26, Stayed the Same | 13
  Week 52, Improved: number analyzed (Participants) | 43
  Week 52, Improved | 30
  Week 52, Worsened: number analyzed (Participants) | 12
  Week 52, Worsened | 2
  Week 52, Stayed the Same: number analyzed (Participants) | 43
  Week 52, Stayed the Same | 11

7. Secondary Outcome: Change From Baseline In Platelet Count At Weeks 26 and 52
Description: The hematologic TMA parameter of platelet count was summarized at baseline and at Week 26 and Week 52 using descriptive statistics for continuous variables for the change from baseline. Results are reported in platelets*10^9/liter (L) blood.
Time Frame: Baseline, Week 26 and Week 52
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of ravulizumab, had at least 1 post-baseline efficacy assessment, met pre-specified eligibility criteria, and had evaluable data at the specified timepoints (Week 26 or 52).
Measure: Median (Full Range); unit: platelets*10^9/L
Arm/Group | Ravulizumab
Number analyzed (Participants) | 56
platelets*10^9/L
  Baseline | 95.25 [18 to 473]
  Change From Baseline at Week 26: number analyzed (Participants) | 48
  Change From Baseline at Week 26 | 125.00 [-126 to 338]
  Change From Baseline at Week 52: number analyzed (Participants) | 44
  Change From Baseline at Week 52 | 126.25 [-51.5 to 335]

8. Secondary Outcome: Change From Baseline In LDH At Weeks 26 and 52
Description: The hematologic TMA parameter of serum LDH was summarized at baseline and at Week 26 and Week 52 using descriptive statistics for continuous variables for the change from baseline. Results are reported in units (U)/L.
Time Frame: Baseline, Week 26 and Week 52
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of ravulizumab, had at least 1 post-baseline efficacy assessment, met pre-specified eligibility criteria, and had evaluable data at the specified timepoints (Week 26 or Week 52).
Measure: Median (Full Range); unit: U/L
Arm/Group | Ravulizumab
Number analyzed (Participants) | 56
U/L
  Baseline | 508.00 [229.5 to 3249]
  Change From Baseline at Week 26: number analyzed (Participants) | 48
  Change From Baseline at Week 26 | -310.75 [-3072 to 8.5]
  Change From Baseline at Week 52: number analyzed (Participants) | 44
  Change From Baseline at Week 52 | -293.75 [-3107 to 81]

9. Secondary Outcome: Change From Baseline In Hemoglobin At Weeks 26 and 52
Description: The hematologic TMA parameter of hemoglobin level was summarized at baseline and at Week 26 and Week 52 using descriptive statistics for continuous variables for the change from baseline. Results are reported in grams (g)/L.
Time Frame: Baseline, Week 26 and Week 52
Population: as for outcome 8
Measure: Median (Full Range); unit: g/L
Arm/Group | Ravulizumab
Number analyzed (Participants) | 56
g/L
  Baseline | 85.00 [60.5 to 140]
  Change From Baseline at Week 26 | 35.00 [-9 to 69]
  Change From Baseline at Week 52: number analyzed (Participants) | 44
  Change From Baseline at Week 52 | 41.75 [-25 to 83.5]

10. Secondary Outcome: Percentage Of Complement Inhibitor Treatment-naïve Participants With An Increase From Baseline In Hemoglobin ≥20 g/L Through Week 26 and Week 52
Description: The percentage of participants with an increase from baseline in hemoglobin ≥20 g/L, observed at 2 separate assessments obtained at least 4 weeks (28 days) apart, and any measurement in between, was assessed through Week 26 and Week 52 and is presented as the percentage of responders, along with a 2-sided 95% CI. The 95% CIs are based on exact confidence limits using the Clopper-Pearson method. To be considered a responder during the 26-week and 52-week Extension Periods, the latest time point a participant could first meet the response criteria was 28 days before the respective Week 26 and Week 52 assessments (components of the response maintained for at least 28 days).
Time Frame: Baseline through Week 26 and through Week 52
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of ravulizumab, had at least 1 post-baseline efficacy assessment, met pre-specified eligibility criteria, and had evaluable data at the specified timepoints (Week 26 or Week 52). Here, Overall Number of Participants analyzed signifies those who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ravulizumab
Number analyzed (Participants) | 38
percentage of participants
  Week 26 | 75.5 [61.1 to 86.7]
  Week 52 | 86.4 [72.6 to 94.8]

11. Secondary Outcome: Change From Baseline In Quality Of Life As Measured By The EuroQol 5-Dimension 3-Level (EQ-5D-3L) At Weeks 26 and 52
Description: The EQ-5D-3L is a participant-answered questionnaire that scores 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression (scored as a 1, 2, or 3, with 3 being the worst health state), as well as health state on a visual analogue scale (0 to 100, with 100 representing the best health state). From these scores, a summary index score is derived using the time trade-off valuation set for the United States and ranges from -1 to 1, where a score above 0.94 indicates full health. An increase in score from baseline indicates improvement in quality of life.
Time Frame: Baseline, Week 26 and Week 52
Population: as for outcome 5
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Ravulizumab
Number analyzed (Participants) | 53
units on a scale
  Baseline | 0.59 [-0.113 to 0.753]
  Change from Baseline at Week 26: number analyzed (Participants) | 46
  Change from Baseline at Week 26 | 0.15 [-0.138 to 0.723]
  Change from Baseline at Week 52: number analyzed (Participants) | 42
  Change from Baseline at Week 52 | 0.26 [-0.143 to 0.707]

12. Secondary Outcome: Change From Baseline In Quality Of Life As Measured By The Functional Assessment Of Chronic Illness Therapy (FACIT)-Fatigue Version 4 Questionnaire At Weeks 26 and 52
Description: Quality of life was evaluated in part using FACIT Fatigue Version 4. The data were summarized at baseline and at the Week 26 and Week 52 time point using descriptive statistics for continuous variables. The FACIT Fatigue Version 4 questionnaire at baseline and the Week 52 timepoint was scored using standard scoring algorithms. The score ranges from 0-52, with a higher score indicating less Fatigue. An increase in score indicated an improvement in quality of life.
Time Frame: Baseline, Week 26 and Week 52
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of ravulizumab, had at least 1 post-baseline efficacy assessment, met pre-specified eligibility criteria, and had evaluable data at the specified timepoints (Week 26 and Week 52).
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Ravulizumab
Number analyzed (Participants) | 48
units on a scale
  Baseline | 24.00 [0 to 51]
  Change From Baseline at Week 26: number analyzed (Participants) | 44
  Change From Baseline at Week 26 | 20.00 [-16 to 48]
  Change From Baseline at Week 52: number analyzed (Participants) | 40
  Change From Baseline at Week 52 | 16.50 [-17 to 50]

ADVERSE EVENTS:
Time Frame: From the beginning of the initial evaluation period (Day1) up to 4.5 years
Arm/Group | Ravulizumab
All-Cause Mortality (participants affected / at risk) | 4/58
Serious Adverse Events (participants affected / at risk) | 38/58
Other Adverse Events (participants affected / at risk) | 56/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ravulizumab (N=58)
Pneumonia (Infections and infestations) | 5 (6)
Septic shock (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (4)
Device related infection (Infections and infestations) | 1 (1)
Escherichia pyelonephritis (Infections and infestations) | 1 (1)
Fungaemia (Infections and infestations) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (3)
Chronic kidney disease (Renal and urinary disorders) | 1 (2)
Hydronephrosis (Renal and urinary disorders) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal haematoma (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Renal pseudoaneurysm (Renal and urinary disorders) | 1 (1)
Atypical haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 2 (2)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (6)
Malignant hypertension (Vascular disorders) | 2 (7)
Hypertensive crisis (Vascular disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (4)
Toothache (Gastrointestinal disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Kidney transplant rejection (Immune system disorders) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Shunt occlusion (Injury, poisoning and procedural complications) | 2 (2)
Biopsy kidney (Investigations) | 2 (2)
Troponin increased (Investigations) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1)
Device leakage (Product Issues) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1)
Nephrectomy (Surgical and medical procedures) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 3 (5)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Peritonitis (Infections and infestations) | 1 (2)
Respiratory tract infection (Infections and infestations) | 1 (1)
Stenotrophomonas infection (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Endophthalmitis (Infections and infestations) | 1 (1)
Enterococcal infection (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Hantaviral infection (Infections and infestations) | 1 (1)
Large intestine infection (Infections and infestations) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Pancreatitis relapsing (Gastrointestinal disorders) | 1 (3)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1)
Shunt stenosis (Injury, poisoning and procedural complications) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Shunt thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Milk allergy (Immune system disorders) | 1 (2)
Transplant rejection (Immune system disorders) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Vitreous disorder (Eye disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ravulizumab (N=58)
Diarrhoea (Gastrointestinal disorders) | 21 (32)
Vomiting (Gastrointestinal disorders) | 17 (22)
Nausea (Gastrointestinal disorders) | 17 (27)
Constipation (Gastrointestinal disorders) | 10 (13)
Abdominal pain (Gastrointestinal disorders) | 6 (9)
Dyspepsia (Gastrointestinal disorders) | 6 (7)
Headache (Nervous system disorders) | 25 (41)
Dizziness (Nervous system disorders) | 7 (7)
Somnolence (Nervous system disorders) | 3 (3)
Urinary tract infection (Infections and infestations) | 12 (25)
Nasopharyngitis (Infections and infestations) | 9 (29)
Oral herpes (Infections and infestations) | 4 (4)
Pyrexia (General disorders) | 13 (14)
Oedema peripheral (General disorders) | 11 (20)
Fatigue (General disorders) | 9 (10)
Pain (General disorders) | 5 (6)
Asthenia (General disorders) | 7 (8)
Face oedema (General disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (17)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (16)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3)
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 (4)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6)
Dry Skin (Skin and subcutaneous tissue disorders) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 7 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 (22)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (10)
Hypertension (Vascular disorders) | 13 (21)
Hypotension (Vascular disorders) | 6 (7)
Contusion (Injury, poisoning and procedural complications) | 3 (5)
Alanine aminotransferase increased (Investigations) | 5 (8)
Aspartate aminotransferase increased (Investigations) | 4 (5)
Anaemia (Blood and lymphatic system disorders) | 10 (10)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
End stage renal disease (Renal and urinary disorders) | 4 (4)
Haematuria (Renal and urinary disorders) | 4 (4)
Anxiety (Psychiatric disorders) | 8 (13)
Insomnia (Psychiatric disorders) | 5 (5)
Vision blurred (Eye disorders) | 4 (5)
Palpitations (Cardiac disorders) | 4 (4)
Drug hypersensitivity (Immune system disorders) | 5 (7)
Abdominal pain upper (Gastrointestinal disorders) | 7 (8)
Gastritis (Gastrointestinal disorders) | 3 (4)
Hypoaesthesia (Nervous system disorders) | 4 (4)
Device related infection (Infections and infestations) | 4 (4)
Gastroenteritis (Infections and infestations) | 4 (4)
Rhinitis (Infections and infestations) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 6 (6)
Catheter site pain (General disorders) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Depression (Psychiatric disorders) | 4 (5)
Haemorrhoids (Gastrointestinal disorders) | 3 (3)
Bronchitis (Infections and infestations) | 5 (5)
Sinusitis (Infections and infestations) | 5 (7)
Pneumonia (Infections and infestations) | 4 (7)
Influenza (Infections and infestations) | 3 (3)
Paraesthesia (Nervous system disorders) | 3 (3)
Presyncope (Nervous system disorders) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Iron deficiency (Metabolism and nutrition disorders) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (4)
Skin abrasion (Injury, poisoning and procedural complications) | 3 (3)
Blood creatinine increased (Investigations) | 3 (3)
Weight decreased (Investigations) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 3 (4)
Dysuria (Renal and urinary disorders) | 3 (3)
Delirium (Psychiatric disorders) | 3 (3)
Intermenstrual bleeding (Reproductive system and breast disorders) | 3 (3)
Ovarian cyst (Reproductive system and breast disorders) | 3 (3)
Cystitis (Infections and infestations) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT02949128/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/28/NCT02949128/SAP_002.pdf